CLINICAL TRIAL: NCT05518968
Title: An Eight-week Program for Family Caregivers of People With Dementia Involving Coach-guided Videoconferencing Sessions With the Use of a Web App Based on Acceptance and Commitment Therapy: A Pilot Study
Brief Title: Videoconferencing Acceptance and Commitment Therapy With a Web App Use for Family Caregivers of People With Dementia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We changed our plan.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Areum Han, Assistant professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300009858
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Depression
Keywords: Acceptance and Commitment Therapy; Alzheimer's Disease; Burden; Caregivers; Dementia; Mindfulness; Self-compassion; Stress; Anxiety; Guilt; Grief; Telemedicine
MeSH Terms: conditions — Depression; Alzheimer Disease; Dementia; Anxiety Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance and Commitment Therapy (Experimental): 8 weekly coach-guided videoconferencing sessions and the use of a web app based on acceptance and commitment therapy
  Interventions: Behavioral: Acceptance and commitment therapy

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — 8 weekly coach-guided videoconferencing sessions and the use of a web app based on acceptance and commitment therapy

SUMMARY:
The purpose of the pilot study is to assess the effects of an 8-week program on improving mental health in depressed family caregivers of people with dementia. The program will involve 8 weekly coach-guided videoconferencing sessions and the use of a web app based on acceptance and commitment therapy (ACT) for 8 weeks. Also, the study aims to understand these caregivers' experiences in the program, including their perspectives on the app features and contents. We aim to recruit 8-10 people for this pilot project. Outcomes regarding caregivers' mental health and ACT processes will be collected at pretest and posttest (after the completion of the 8-week program) and compared over time (i.e., posttest scores compared to pretest). At posttest, acceptability and perceived usability of the app will be evaluated using the 10-item System Usability Scale and 30-40 minute individual interviews.

DETAILED DESCRIPTION:
The purpose of the pilot study is to assess the effects of an 8-week program on improving mental health in depressed family caregivers of people with dementia. The program will involve 8 weekly coach-guided videoconferencing sessions and the use of a web app based on acceptance and commitment therapy (ACT) for 8 weeks. Also, the study aims to understand these caregivers' experiences in the program, including their perspectives on the app features and contents. We aim to recruit 8-10 people for this pilot project. Outcomes regarding caregivers' mental health and ACT processes will be collected at pretest and posttest (after the completion of the 8-week program) and compared over time (i.e., posttest scores compared to pretest). At posttest, acceptability and perceived usability of the app will be evaluated using the 10-item System Usability Scale and 30-40 minute individual interviews. Participants' characteristics will be summarized using descriptive statistics. Either the Wilcoxon signed-rank test (a non-parametric test) or the paired sample t-test (a parametric test) will be performed to test the exploratory hypothesis that participants' scores for the outcome measures would significantly improve at posttest compared to pretest. Because of the exploratory nature of the study, no adjustment of p values will be conducted for multiple statistical comparisons of the outcome measures. Statistical significance will be set at p <.05, and the effect sizes derived from this pilot study will form a basis for determining a sample size with sufficient statistical power required for a subsequent clinical trial. Caregivers' experiences in the app use and perspectives on the developed app will be explored using individual Zoom interviews. Interpretative phenomenological analysis will be used to analyze the interview data.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling adults (age 18 or over) who are currently taking the primary responsibility for the care of a relative with dementia living in the community
* having at least mild depression as measured by the Patient Health Questionnaire (PHQ)-9
* having a web-enabled device (e.g., a smartphone, a tablet, or a laptop/desktop) with the internet access at home

Exclusion Criteria:

* having cognitive, physical, or sensory deficits or language barriers (non-English communicator) that might impede study participation
* receiving a psychological therapy at the time of recruitment
* having a prior experience in acceptance and commitment therapy
* having psychiatric hospitalizations in the previous two years
* considering or planning to place relatives with dementia in a nursing home within 3 months
* recent frequent hospitalizations of their relatives with dementia that might contribute to study dropout

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to immediately after the 8-week intervention on the Patient Health Questionnaire-9 | Change from baseline to immediately after the 8-week intervention
  The Patient Health Questionnaire-9 is a 9-item questionnaire assessing depressive symptoms on a scale of 0 to 3. Scores range from 0 to 27. Higher scores indicate greater symptomatology in depression.

SECONDARY OUTCOMES:
Change from baseline to immediately after the 8-week intervention on the Generalized Anxiety Disorder-7 | Change from baseline to immediately after the 8-week intervention
  The Generalized Anxiety Disorder-7 is a 7-item questionnaire assessing anxiety on a scale of 0 to 3. Scores range from 0 to 21. Higher scores indicate greater anxiety.
Change from baseline to immediately after the 8-week intervention on the Perceived Stress Scale | Change from baseline to immediately after the 8-week intervention
  The Perceived Stress Scale is a 10-item questionnaire assessing stress on a scale of 0 to 4. Scores range from 0 to 40. Higher scores indicate greater stress.
Change from baseline to immediately after the 8-week intervention on the World Health Organization Quality of Life - Psychological health component | Change from baseline to immediately after the 8-week intervention
  World Health Organization Quality of Life - Psychological health component has 6 items measuring psychological quality of life on scale of 1 to 5. Scores range from 6 to 30. Higher scores denote higher quality of life in terms of psychological health.
Change from baseline to immediately after the 8-week intervention on the Zarit Burden Interview | Change from baseline to immediately after the 8-week intervention
  Zarit Burden Interview is a 12-item self-report questionnaire assessing caregiver burden on a scale of 0 to 4. Higher scores indicate higher levels of burden. The total scores range from 0 to 48, and scores of 17 or greater indicate severe/high burden.
Change from baseline to immediately after the 8-week intervention on the Marwit-Meuser Caregiver Grief Inventory Brief-Form | Change from baseline to immediately after the 8-week intervention
  Marwit-Meuser Caregiver Grief Inventory Brief-Form is a 6-item self-report questionnaire assessing grief of caregivers on a scale of 1 to 5. Scores range from 6 to 30. Higher scores indicate higher levels of grief.
Change from baseline to immediately after the 8-week intervention on the Caregiver Guilt Questionnaire | Change from baseline to immediately after the 8-week intervention
  Caregiver Guilt Questionnaire is a 22-item self-report questionnaire assessing feelings of guilt in caregivers on a scale of 0 to 4. Scores range from 0 to 88. Higher scores indicate higher levels of guilt.
Change from baseline to immediately after the 8-week intervention on the Self-Compassion Scale-Short Form | Change from baseline to immediately after the 8-week intervention
  Self-Compassion Scale- Short Form is a 12-item self-report questionnaire assessing self-compassion on a scale of 1 to 5. Scores range from 12 to 60. Higher scores indicate higher levels of self-compassion.
Change from baseline to immediately after the 8-week intervention on the Action and Acceptance Questionnaire-II | Change from baseline to immediately after the 8-week intervention
  Action and Acceptance Questionnaire -II is a 7-item self-report questionnaire measuring psychological flexibility on a scale of 1 to 7. Scores range from 7 to 49. Higher scores indicate poor psychological flexibility.
Change from baseline to immediately after the 8-week intervention on the Cognitive Fusion Questionnaire | Change from baseline to immediately after the 8-week intervention
  Cognitive Fusion Questionnaire -7 is a 7-item self-report questionnaire measuring cognitive fusion on scale of 1 to 7. Scores range from 7 to 49. Higher scores indicate greater levels of cognitive fusion.
Change from baseline to immediately after the 8-week intervention on the Engaged Living Scale | Change from baseline to immediately after the 8-week intervention
  Engaged Living Scale -9 is a 9-item self-assessment instrument that measures clarity and engagement with personal values and life fulfillment on a scale of 1 to 5. The total scores range from 9 to 45, and higher scores indicate increased clarity and engagement with personal values and greater life fulfillment.
Change from baseline to immediately after the 8-week intervention on the Five Facet Mindfulness Questionnaire | Change from baseline to immediately after the 8-week intervention
  Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item self-assessment instrument that measures five aspects of mindfulness (i.e., observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience) on a scale of 1 to 5. The total scores range from 39 to 195, and higher scores indicate greater mindfulness.

OTHER OUTCOMES:
System Usability Scale | immediately after the 8-week intervention
  The System Usability Scale (SUS) is a 10-item self-report questionnaire measuring usability of a tool/program/intervention. Higher scores indicate greater levels of perceived usability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Areum Han, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No